CLINICAL TRIAL: NCT04214028
Title: Real World Evidence of the Safety and Clinical Practice Use of Maviret in Adolescents Patients Infected With Chronic Hepatitis C Virus (All Case Survey)
Brief Title: A Study of the Safety, Effectiveness and Clinical Use of Maviret in Adolescent Patients With Chronic Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-620
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Hepatitis C Virus (HCV); Chronic Hepatitis C (CHC); Maviret; Mavyret
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Maviret Participants: Participants receiving glecaprevir plus pibrentasvir (GLE/PIB, other names: Maviret) as routine standard of care for HCV.

SUMMARY:
This study will assess the safety and effectiveness of Maviret (Glecaprevir plus Pibrentasvir (GLE/PIB)) in adolescent participants diagnosed with chronic hepatitis C (CHC) in a real world setting across clinical practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Hepatitis C Virus (HCV) infection treated in daily practice with Maviret
* Enrolled after Maviret treatment begins
* Prior treatment with Maviret

Exclusion Criteria:

None

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants aged ≥ 12 to <18 years of age with chronic hepatitis C receiving Maviret in accordance with local label.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Drug Reactions (ADRs) | Up to approximately 36 weeks
  Adverse drug reactions are defined as adverse events of which a causal relationship with Maviret could not be ruled out.
Percentage of Participants with Adverse Drug Reactions (ADRs) | Up to approximately 36 weeks
  Adverse drug reactions are defined as adverse events of which a causal relationship with Maviret could not be ruled out.
Number of Participants with Serious Adverse Events (SAEs) | Up to approximately 36 weeks
  A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgement, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent serious adverse events (TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to approximately 36 weeks
  A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgement, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent serious adverse events (TESAEs) are defined as any event that began or worsened in severity after the first dose of study drug.

SECONDARY OUTCOMES:
Percentage of participants achieving Sustained Virologic Response 12 (SVR12) | At Week 12
  Defined as HCV Ribonucleic acid (RNA) not detected 12 weeks after the last dose of study drug.
Percentage of participants achieving Sustained Virologic Response (SVR) | At 4, 8, 12 and 24 weeks after last dose of Maviret (up to approximately 36 weeks)
  SVR defined as HCV Ribonucleic acid (RNA) < Lower limit of quantification (LLOQ).
Percentage of Participants with On-Treatment Virologic Failure (Breakthrough) | Up to approximately 36 weeks
  On-treatment virologic failure (breakthrough) defined as at least 1 documented HCV RNA < 50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment or failure to suppress (each measured on-treatment HCV RNA value ≥ 50 IU/mL).
Percentage of Participants with After-Treatment Virologic Failure (Relapse) | Up to approximately 36 weeks
  After-treatment virologic failure (relapse) is defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 24 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (54):
- Japan (54):
  - Kariya Toyota General Hospital /ID# 239046, Kariya-shi, Aichi-ken
  - Meijo Hospital /ID# 250955, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 226746, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 238745, Nagoya, Aichi-ken
  - Hirosaki University Hospital /ID# 262654, Hirosaki-shi, Aomori
  - Misawa Municipal Misawa Hospital /ID# 229544, Misawa-shi, Aomori
  - Chiba University Hospital /ID# 225889, Chiba, Chiba
  - Japanese Red Cross Narita Hospital /ID# 261349, Narita-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 239387, Matsuyama, Ehime
  - Shikoku Central Hospital of the Mutual Aid /ID# 230273, Shikokuchūō, Ehime
  - Kyushu University Hospital /ID# 261351, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 255088, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital /ID# 224112, Kurume-shi, Fukuoka
  - Aoyama Clinic /ID# 261942, Koriyama-shi, Fukushima
  - Shirakawa Kosei General Hosp. /ID# 240816, Shirakawa-shi, Fukushima
  - Gifu Municipal Hospital /ID# 225890, Gifu, Gifu
  - Machida Clinic /ID# 238744, Maebashi, Gunma
  - Gunma University Hospital /ID# 231700, Maebashi, Gunma
  - Heisei Hidaka Clinic /ID# 231758, Takasaki, Gunma
  - Kousei General Hospital /ID# 249395, Mihara-shi, Hiroshima
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 239388, Amagasaki-shi, Hyōgo
  - Hyogo Prefectural Amagasaki General Medical Center /ID# 261350, Amagasaki-shi, Hyōgo
  - Fujikawa Clinic /ID# 221135, Kanzaki-gun, Hyōgo
  - Takano Kids Clinic /ID# 251656, Kobe, Hyōgo
  - University of tsukuba Hospital /ID# 267373, Tsukuba, Ibaraki
  - Yamada Clinic /ID# 225909, Fujisawa-shi, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 221136, Sagamihara-shi, Kanagawa
  - Kawaguchi Clinic /ID# 226843, Yokohama, Kanagawa
  - Kumamoto Shinto General Hospital /ID# 223245, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine /ID# 229599, Kyoto, Kyoto
  - Kyoto Shimogamo Hospital /ID# 233903, Kyoto, Kyoto
  - Okanami General Hospital /ID# 256995, Iga-shi, Mie-ken
  - Ise Red Cross Hospital /ID# 222018, Ise-shi, Mie-ken
  - Mie University Hospital /ID# 233864, Tsu, Mie-ken
  - Miyagi Children's Hospital /ID# 258143, Sendai, Miyagi
  - Aizawa Hospital /ID# 223247, Matsumoto-shi, Nagano
  - Nara Hospital Kinki University Faculty of Medicine, /ID# 224609, Ikoma-shi, Nara
  - Nakatsu Municipal Hospital /ID# 233390, Nakatsu-shi, Oita Prefecture
  - Watanabe Clinic /ID# 261352, Kasaoka-shi, Okayama-ken
  - Heartlife Hospital /ID# 249394, Nakagami-gun, Okinawa
  - Kitano Hospital /ID# 255150, Osaka, Osaka
  - Yumura Clinic /ID# 254478, Osaka, Osaka
  - Osaka University Hospital /ID# 256174, Suita-shi, Osaka
  - Saitama Medical University Hospital /ID# 258144, Iruma-gun, Saitama
  - Saitama Children's Medical Center /ID# 227633, Saitama-shi, Saitama
  - Tsukada Clinic /ID# 255152, Maibara-shi, Shiga
  - Tamakoshi Clinic /ID# 224113, Hamamatsu, Shizuoka
  - Tokyo Metropolitan Children's Medical Center /ID# 258142, Fuchu-shi, Tokyo
  - National Center for Child Health and Development /ID# 225293, Setagaya-ku, Tokyo
  - Tottori University Hospital /ID# 227634, Yonago-shi, Tottori
  - Ishibashi Clinic /ID# 258148, Yonezawa-shi, Yamagata
  - Yamaguchi University Hospital /ID# 262655, Ube-shi, Yamaguchi
  - Oita Cardiovascular Hospital /ID# 239725, Ōita
  - Shonai Hospital /ID# 232294, Yamagata

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P19-620#additional-resources-section